CLINICAL TRIAL: NCT06561048
Title: A Phase 3, Randomized, Open-Label Study to Investigate the Efficacy and Safety of ITK Inhibitor Soquelitinib Versus Physician's Choice Standard of Care Treatment (Selected Single Agent) in Participants With Relapsed/Refractory Peripheral T-cell Lymphoma Not Otherwise Specified, Follicular Helper T-cell Lymphomas, or Systemic Anaplastic Large-cell Lymphoma
Brief Title: Soquelitinib vs Standard of Care in Participants With Relapsed/Refractory Peripheral T-cell Lymphoma Not Otherwise Specified, Follicular Helper T-cell Lymphomas, or Systemic Anaplastic Large-cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Corvus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPI-818-004
Record Dates: First submitted 2024-08-16; First posted 2024-08-19 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Peripheral T-Cell Lymphoma, Not Otherwise Specified; Angioimmunoblastic T-cell Lymphoma; Follicular T-Cell Lymphoma; Nodal Peripheral T-Cell Lymphoma With TFH Phenotype; Systemic Anaplastic Large Cell Lymphoma; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell
Keywords: Peripheral T-Cell Lymphoma, Not Otherwise Specified (PTCL-NOS); Follicular Helper T-Cell Lymphoma (FHTCL); Angioimmunoblastic T-cell Lymphoma (AITL); Follicular T-Cell Lymphoma (FTCL); Nodal Peripheral T-Cell Lymphoma with T Follicular Helper Phenotype (PTCL-Tfh); Systemic Anaplastic Large Cell Lymphoma (sALCL)
MeSH Terms: conditions — Lymphoma, T-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell, Peripheral | interventions — belinostat; 10-propargyl-10-deazaaminopterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Soquelitinib (Experimental): Participants will administer soquelitinib 200 mg orally twice daily for up to 2 years
  Interventions: Drug: Soquelitinib
- Standard of Care (Active Comparator): Participants will receive physician's choice standard of care treatment of either pralatrexate or belinostat for up to 2 years
  Interventions: Drug: Belinostat; Drug: Pralatrexate

INTERVENTIONS:
Drug: Soquelitinib — Soquelitinib 200 mg tablets will be taken by mouth two times a day
  Other Names: CPI-818
  Arms: Soquelitinib
Drug: Belinostat — Belinostat (1000 mg/m2) will be administered by intravenous infusion once daily on Days 1 through 5 of each 21-day cycle
  Other Names: Beleodaq®
  Arms: Standard of Care
Drug: Pralatrexate — Pralatrexate (30 mg/m2) will be administered intravenously over 3 to 5 minutes once weekly for 6 weeks in each 7-week cycle
  Other Names: Folotyn®
  Arms: Standard of Care

SUMMARY:
A Phase 3, randomized, 2-arm, open-label, multicenter, stratified study of soquelitinib versus physician's choice standard of care (SOC) treatment (selected single agents) in participants with relapsed/refractory (R/R) peripheral T-cell lymphoma not otherwise specified (PTCL-NOS), follicular helper T-cell lymphomas (FHTCLs), or systemic anaplastic large-cell lymphoma (sALCL).

DETAILED DESCRIPTION:
This is a Phase 3, randomized, 2-arm, open-label, multicenter, stratified study of soquelitinib, an oral interleukin-2-inducible T cell kinase (ITK) inhibitor, versus physician's choice standard of care (SOC) treatment of either belinostat or pralatrexate in participants with relapsed/refractory (R/R) peripheral T-cell lymphoma not otherwise specified (PTCL-NOS), follicular helper T-cell lymphomas (FHTCLs), or systemic anaplastic large-cell lymphoma (sALCL). Approximately 150 participants will be randomized at a 1:1 ratio to the 2 treatment arms (soquelitinib or SOC) and will be stratified by region of the world, age, and time to relapse for the most recent prior therapy. Participants will receive study treatment for up to a maximum of 2 years, unacceptable toxicity, or disease progression, whichever is earlier. Participants randomized to receive SOC who have confirmation of progressive disease may have the opportunity to crossover to receive treatment with soquelitinib.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants ≥18 years of age on the day of signing the informed consent form.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
3. Histologically confirmed PTCL-NOS, FHTCLs or sALCL per The International Consensus Classification of Mature Lymphoid Neoplasms.
4. Progressed on, be refractory to, relapsed, or intolerant to standard therapy for their cancer. At least 1 but not more than 3 prior systemic therapies.
5. Fluorodeoxyglucose-avid disease by positron emission tomography and measurable disease of at least 1.5 cm by computed tomography, as assessed by the site radiologist.
6. Life expectancy >12 weeks.
7. Adequate organ function as determined by:

   * Absolute neutrophil count ≥ 1.0×10^9/L (1000/mm3) (without receiving granulocyte-colony stimulating factor)
   * Platelet count ≥ 100×10^9/L (without transfusion)
   * Hemoglobin ≥ 9.0 g/dL, without packed red blood cell transfusion within the last 1 week of starting study drug
   * Prothrombin time international normalized ratio and partial thromboplastin time ≤1.5 × upper limit of normal (ULN), unless participant is receiving anticoagulant therapy and prothrombin time or activated partial thromboplastin time is within therapeutic range of intended use of anticoagulants
   * Calculated creatinine clearance (CrCl) according to Cockcroft-Gault formula and based on ideal body weight or 24-hour urine CrCl ≥ 50 mL/minute
   * Total bilirubin ≤ 1.5 × ULN or direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 × ULN. For participants with Gilbert's disease: ≤ 3.0 mg/dL or discussion with the Medical Monitor
   * Aspartate aminotransferase and alanine transaminase ≤ 2.5 × ULN (≤ 5 × ULN for participants with liver metastases)
   * Serum albumin > 2.5 g/dL
   * Serum calcium < 12 mg/dL or corrected serum calcium < ULN
8. Must have recovered from all AEs due to previous therapies to Grade ≤ 1 or baseline except for the following:

   * Grade ≤ 2 neuropathy
   * Alopecia and non-acute toxicities
   * If major received major surgery, then must have recovered adequately per the investigator from the toxicity and/or complications from the intervention prior to starting study treatment
9. Female participants of childbearing potential who are sexually active with a non-sterilized male partner must agree to use at least 1 highly effective method of contraception from the time of screening and must agree to continue using such precautions for 120 days after the last dose of study drug for participants who receive soquelitinib, or 6 months after the last dose for participants who receive either belinostat or pralatrexate.
10. Non-sterilized males who are sexually active with a female partner of childbearing potential must use a condom plus spermicide from Day 1 through 120 days after the last dose of study drug.

Exclusion Criteria:

1. Participants who have T-cell lymphoma with active central nervous system involvement.
2. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study.
3. History of primary immunodeficiency or sold organ transplantation.
4. History of opportunistic infection within 30days of screening requiring active systemic treatment or active infection requiring IV therapy.
5. Any active infection requiring IV therapy.
6. History of invasive prior malignancy that required systemic therapy within last 3 years.
7. Any condition that confounds the ability to interpret data from the study.
8. Known to be positive for HIV, or positive test for chronic hepatitis B virus (HBV) infection (defined as positive hepatitis B surface antigen [HBsAg]) or positive test for hepatitis C antibody.
9. Monoclonal antibody therapy for cancer, radiotherapy, or chemotherapy within 3 weeks and targeted therapy within 2 weeks prior to the first dose of study treatment.
10. Prior administration of an ITK inhibitor.
11. Participants who need immediate cytoreductive therapy.
12. Participants requiring the concomitant use of strong inhibitors or inducers of CYP3A or who have received these within 5 half-lives or 14 days prior to the start of study treatment.
13. History of allogeneic hematopoietic stem cell transplantation.
14. Candidate for hematopoietic stem cell transplantation at screening.
15. History of progressive disease within 6 months of autologous hematopoietic stem cell transplantation.
16. Concurrent enrollment in another clinical study
17. Females who are pregnant, lactating, or intend to become pregnant during their participation in the study, starting with the screening visit through 6 months after the last dose of study treatment.
18. Participants who cannot ingest medications orally or who have malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to 4 years post study treatment initiation
  Time from first study treatment to first occurrence of progression (as assessed by the Independent Review Committee) or death, whichever occurs first

SECONDARY OUTCOMES:
Objective response rate | Up to 2 years post study treatment initiation
  The rate of participants who achieve a partial response or complete response as assessed by the Independent Review Committee according to the Revised Criteria for Response Assessment of Malignant Lymphoma (Lugano Classification 2014), and modified Severity Weighted Assessment Tool (mSWAT) for participants with skin involvement
Overall survival | Up to 4 years post study treatment initiation
  Time from first study treatment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Mahabhashyam, MD, MPH, Study Director — Corvus Pharmaceuticals, Inc.
Locations (1):
- Corvus Pharmaceuticals, South San Francisco, California, United States